CLINICAL TRIAL: NCT00065806
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Test the Safety and Efficacy of Lipitor (Atorvastatin) in Reducing the Progression of Carotid IMT in Early Childhood SLE
Brief Title: Atherosclerosis Prevention in Pediatric Lupus Erythematosus (APPLE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laura Schanberg (Other)
Responsible Party: Sponsor-Investigator, Laura Schanberg, Associate Director, Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00006680; NIAMS-090; N01AR022265 (NIH)
Record Dates: First submitted 2003-08-01; First posted 2003-08-04 (Estimated); Results first posted 2013-08-15 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-07

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Pediatric lupus; Atherosclerosis; SLE; HMG CoA reductase inhibitor
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Atherosclerosis | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients will be treated with dietary intervention (AHA Therapeutic Lifestyle Changes [TLC] diet, [http://www.nhlbi.nih.gov/cgi-bin/chd/step2intro.cgi]), cardiovascular risk factor reduction counseling, hydroxychloroquine, low-dose aspirin, a multivitamin containing folate, plus atorvastatin at 10 mg or 20 mg depending on the patient's weight. Patients weighing more than 50 kg will receive 10 mg qd atorvastatin for the first month, which will be increased to 20 mg qd at the Day 30 visit and continue through month 36. Participants weighing less than 50kg will receive a maximum of 10 mg po qd for 36 months.
  Interventions: Drug: Atorvastatin
- 2 (Placebo Comparator): Patients will be treated with dietary intervention (AHA Therapeutic Lifestyle Changes [TLC] diet, [http://www.nhlbi.nih.gov/cgi-bin/chd/step2intro.cgi]), cardiovascular risk factor reduction counseling, hydroxychloroquine, low-dose aspirin, a multivitamin containing folate, plus placebo at 10 mg or 20 mg depending on the patient's weight. Patients weighing more than 50 kg will receive 10 mg qd placebo for the first month, which will be increased to 20 mg qd at the Day 30 visit and continue through month 36. Participants weighing less than 50kg will receive a maximum of 10 mg po qd for 36 months.
  Interventions: Drug: Placebo atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Participants weighing more 50 kg will receive 10 mg of atorvastatin po qd as a starting dose, which will be increased to 20 mg po qd at the Day 30 visit and continue through month 36. Participants weighing less than 50 kg will receive a maximum of 10 mg po qd for 36 months.
  Other Names: Lipitor; Atorvastatin Calcium
  Arms: 1
Drug: Placebo atorvastatin — Participants weighing more 50 kg will receive 10 mg of placebo po qd as a starting dose, which will be increased to 20 mg po qd at the Day 30 visit and continue through month 36. Participants weighing less than 50 kg will receive a maximum of 10 mg po qd for 36 months.
  Arms: 2

SUMMARY:
The purpose of this study is:

1. To assess the efficacy of a lipid-lowering agent (atorvastatin) on the development of atherosclerosis that predisposes children with SLE to cardiovascular events in adulthood.
2. To assess the safety of intermediate-term (36 months) treatment of children and young adults with atorvastatin.
3. To further characterize the course of SLE in children and young adults, by establishing a cohort of pediatric SLE patients to be followed prospectively.
4. To establish a mechanism for conducting clinical trials in rare pediatric rheumatic diseases using the Children's Arthritis and Rheumatology Research Alliance (CARRA).

DETAILED DESCRIPTION:
Children and adolescents with SLE represent 15% of all SLE patients. Children with SLE suffer high morbidity that affects many organ systems, reduces their quality of life, and shortens their lifespan. As more children with SLE survive into adulthood, atherosclerotic cardiovascular disease has emerged as a major concern. SLE is a significant risk factor for myocardial infarction and death in young premenopausal women with SLE, even after controlling for traditional cardiovascular risk factors. Acceleration of atherogenesis in SLE most likely reflects SLE-associated vascular immune and inflammatory changes.

Although limited, the data on cardiovascular and lipid abnormalities in children with SLE implicate atherosclerosis as an important cause of long-term morbidity and mortality. The 3-hydroxy-3-methlglutaryl-coenzyme A (HMG CoA) reductase inhibitors, or statins, reduce mortality and morbidity from atherosclerosis in adults and have intrinsic anti-inflammatory and immune modulatory properties. These anti-inflammatory and immune modulatory activities may have particular benefit in the prevention and treatment of atherosclerosis in SLE. This trial will evaluate atorvastatin in children with SLE in the largest cohort of pediatric SLE patients ever studied prospectively.

Children in this study will be randomized to receive either atorvastatin or a placebo. All children will be followed for 3 years, during which they will have 15 study visits. Study visits will generally last 2 hours and will include medical interview, medication review and pill count, physical examination, and blood and urine tests. Cardiovascular-specific outcome measures will include assessments of high sensitivity CRP; fasting lipid profile; homocysteine level; apolipoprotein A, B1, and Lp(a); carotid intima media thickness (IMT); and tensor diffusion/MRI.

ELIGIBILITY:
Inclusion Criteria:

* Meets American College of Rheumatology (ACR) revised diagnostic guidelines for SLE
* Weight of 25 kg (55 lbs) or more
* Outpatient
* Ability to complete self-report questionnaires in either English or Spanish
* Willingness to comply with recommended diet
* Acceptable methods of contraception

Exclusion Criteria:

* Drug-induced lupus
* Liver disease (ALT or aspartate aminotransferase greater than 2 X normal value)
* Myositis (CK greater than 3 X normal value)
* Inability to obtain adequate-quality IMT images
* Current use of oral or parenteral tacrolimus or cyclosporine
* Dialysis or serum creatinine reater than 2.5 mg/dL
* Active nephrotic syndrome (urinary protein greater than 3 g/24 h and serum albumin less than 2.3 g/dl)
* Total cholesterol greater than 350 mg/dL
* Xanthoma
* Familial hypercholesterolemia
* Pregnant or breastfeeding
* Use of estrogen-containing contraceptives (e.g., Lo-Ovral)
* Unable to adhere to study regimen
* Life-threatening non-SLE illness that would interfere with ability to complete the study
* Current drug or alcohol abuse
* Anticipated poor compliance
* Participation in another drug intervention study within 30 days of study enrollment

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 221 (Actual)
Dates: Start 2003-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura E. Schanberg, MD, Principal Investigator — Duke Medical Center
Locations (1):
- Duke Medical Center / Duke Clinical Research Institute, Durham, North Carolina, United States

REFERENCES:
- [Derived] Gurion R, Tangpricha V, Yow E, Schanberg LE, McComsey GA, Robinson AB; Atherosclerosis Prevention in Pediatric Lupus Erythematosus Investigators. Avascular necrosis in pediatric systemic lupus erythematosus: a brief report and review of the literature. Pediatr Rheumatol Online J. 2015 Apr 23;13:13. doi: 10.1186/s12969-015-0008-x. PMID 25902709
- [Derived] Robinson AB, Tangpricha V, Yow E, Gurion R, Schanberg LE, McComsey GA; APPLE Investigators. Vitamin D status is a determinant of atorvastatin effect on carotid intima medial thickening progression rate in children with lupus: an Atherosclerosis Prevention in Pediatric Lupus Erythematosus (APPLE) substudy. Lupus Sci Med. 2014 Sep 10;1(1):e000037. doi: 10.1136/lupus-2014-000037. eCollection 2014. PMID 25396067
- [Derived] Robinson AB, Tangpricha V, Yow E, Gurion R, McComsey GA, Schanberg LE; APPLE Investigators. Vitamin D deficiency is common and associated with increased C-reactive protein in children and young adults with lupus: an Atherosclerosis Prevention in Pediatric Lupus Erythematosus substudy. Lupus Sci Med. 2014 Apr 30;1(1):e000011. doi: 10.1136/lupus-2014-000011. eCollection 2014. PMID 25396060
- [Derived] Ardoin SP, Schanberg LE, Sandborg CI, Barnhart HX, Evans GW, Yow E, Mieszkalski KL, Ilowite NT, Eberhard A, Imundo LF, Kimura Y, Levy D, von Scheven E, Silverman E, Bowyer SL, Punaro L, Singer NG, Sherry DD, McCurdy DK, Klein-Gitelman M, Wallace C, Silver RM, Wagner-Weiner L, Higgins GC, Brunner HI, Jung L, Soep JB, Reed AM, Thompson SD; APPLE investigators. Secondary analysis of APPLE study suggests atorvastatin may reduce atherosclerosis progression in pubertal lupus patients with higher C reactive protein. Ann Rheum Dis. 2014 Mar;73(3):557-66. doi: 10.1136/annrheumdis-2012-202315. Epub 2013 Feb 22. PMID 23436914
- [Derived] Schanberg LE, Sandborg C, Barnhart HX, Ardoin SP, Yow E, Evans GW, Mieszkalski KL, Ilowite NT, Eberhard A, Imundo LF, Kimura Y, von Scheven E, Silverman E, Bowyer SL, Punaro M, Singer NG, Sherry DD, McCurdy D, Klein-Gitelman M, Wallace C, Silver R, Wagner-Weiner L, Higgins GC, Brunner HI, Jung L, Soep JB, Reed AM, Provenzale J, Thompson SD; Atherosclerosis Prevention in Pediatric Lupus Erythematosus Investigators. Use of atorvastatin in systemic lupus erythematosus in children and adolescents. Arthritis Rheum. 2012 Jan;64(1):285-96. doi: 10.1002/art.30645. PMID 22031171
- [Derived] Schanberg LE, Sandborg C, Barnhart HX, Ardoin SP, Yow E, Evans GW, Mieszkalski KL, Ilowite NT, Eberhard A, Levy DM, Kimura Y, von Scheven E, Silverman E, Bowyer SL, Punaro L, Singer NG, Sherry DD, McCurdy D, Klein-Gitelman M, Wallace C, Silver R, Wagner-Weiner L, Higgins GC, Brunner HI, Jung L, Soep JB, Reed A; Atherosclerosis Prevention in Pediatric Lupus Erythematosus Investigators. Premature atherosclerosis in pediatric systemic lupus erythematosus: risk factors for increased carotid intima-media thickness in the atherosclerosis prevention in pediatric lupus erythematosus cohort. Arthritis Rheum. 2009 May;60(5):1496-507. doi: 10.1002/art.24469. PMID 19404953

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 Atorvastatin: Patients will be treated with dietary intervention (AHA Therapeutic Lifestyle Changes [TLC] diet, [http://www.nhlbi.nih.gov/cgi-bin/chd/step2intro.cgi]), cardiovascular risk factor reduction counseling, hydroxychloroquine, low-dose aspirin, a multivitamin containing folate, plus atorvastatin at 10 mg or 20 mg depending on the patient's weight. Patients weighing more than 50 kg will receive 10 mg qd atorvastatin for the first month, which will be increased to 20 mg qd at the Day 30 visit and continue through month 36. Participants weighing less than 50kg will receive a maximum of 10 mg po qd for 36 months.
  Atorvastatin : Participants weighing more 50 kg will receive 10 mg of atorvastatin po qd as a starting dose, which will be increased to 20 mg po qd at the Day 30 visit and continue through month 36. Participants weighing less than 50 kg will receive a maximum of 10 mg po qd for 36 months.
- 2 Placebo: Patients will be treated with dietary intervention (AHA Therapeutic Lifestyle Changes [TLC] diet, [http://www.nhlbi.nih.gov/cgi-bin/chd/step2intro.cgi]), cardiovascular risk factor reduction counseling, hydroxychloroquine, low-dose aspirin, a multivitamin containing folate, plus placebo at 10 mg or 20 mg depending on the patient's weight. Patients weighing more than 50 kg will receive 10 mg qd placebo for the first month, which will be increased to 20 mg qd at the Day 30 visit and continue through month 36. Participants weighing less than 50kg will receive a maximum of 10 mg po qd for 36 months.
  Placebo atorvastatin : Participants weighing more 50 kg will receive 10 mg of placebo po qd as a starting dose, which will be increased to 20 mg po qd at the Day 30 visit and continue through month 36. Participants weighing less than 50 kg will receive a maximum of 10 mg po qd for 36 months.
Period: Overall Study
Arm/Group | 1 Atorvastatin | 2 Placebo
Started | 113 | 108
Completed | 93 | 89
Not Completed | 20 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Atorvastatin | 2 Placebo | Total
Number analyzed (Participants) | 113 | 108 | 221
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 87 | 87 | 174
  Between 18 and 65 years | 26 | 21 | 47
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 15.7 (2.8) | 15.8 (2.5) | 15.7 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 89 | 184
  Male | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean-Mean Common Carotid IMT (CIMT)
Description: For the common carotid arterial segment, mean CIMT values were averaged across angles by side and wall to produce 4 summary variables (right common near wall mean, right common far wall mean, left common near wall mean and left common far wall mean). These summary variables were then averaged to estimate a single mean-mean common CIMT for each participant visit.
Time Frame: Change from baseline to 36 months
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | 1 Atorvastatin | 2 Placebo
Number analyzed (Participants) | 113 | 108
mm | 0.0010 [-0.0006 to 0.0026] | 0.0024 [0.0007 to 0.0040]

2. Secondary Outcome: Change in Mean-Max CIMT
Description: For each side, segment and wall, the maximum CIMT over the 4 angles of interrogation was selected to produce 12 summary variables (right common near wall max, right common far wall max, right bifurcation near wall max, right bifurcation far wall max, right internal near wall max, right internal far wall max, left common near wall max, left common far wall max, left bifurcation near wall max, left bifurcation far wall max, left internal near wall max and left internal far wall max). These 12 summary variables were then averaged to estimate a single mean-max CIMT for each participant visit.
Time Frame: Change from baseline to 36 months
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | 1 Atorvastatin | 2 Placebo
Number analyzed (Participants) | 113 | 108
mm | 0.0037 [0.0015 to 0.0058] | 0.0064 [0.0042 to 0.0086]

3. Secondary Outcome: Change in Mean-Mean CIMT
Description: For each side, segment and wall, mean CIMT values were averaged over the 4 angles of interrogation to produce 12 summary variables (right common near wall mean, right common far wall mean, right bifurcation near wall mean, right bifurcation far wall mean, right internal near wall mean, right internal far wall mean, left common near wall mean, left common far wall mean, left bifurcation near wall mean, left bifurcation far wall mean, left internal near wall mean and left internal far wall mean). These 12 summary variables were then averaged to estimate a single mean-mean CIMT for each participant visit.
Time Frame: Change from baseline to 36 months
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | 1 Atorvastatin | 2 Placebo
Number analyzed (Participants) | 113 | 108
mm | 0.0033 [0.0018 to 0.0047] | 0.0049 [-0.0034 to 0.0063]

4. Secondary Outcome: Change in Mean-Max Common CIMT
Description: For each side and wall of the common carotid arterial segment, the maximum CIMT over the 4 angles of interrogation was selected to produce 4 summary variables (right common near wall max, right common far wall max, left common near wall max and left common far wall max). These summary variables were then averaged to estimate a single mean-max common CIMT for each participant visit.
Time Frame: Change from baseline to 36 months
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | 1 Atorvastatin | 2 Placebo
Number analyzed (Participants) | 113 | 108
mm | 0.0006 [-0.0018 to 0.003] | 0.0008 [-0.0017 to 0.003]

5. Secondary Outcome: Change in Mean-Max Internal CIMT
Description: For each side and wall of the internal carotid arterial segment, the maximum CIMT over the 4 angles of interrogation was selected to produce 4 summary variables (right internal near wall max, right internal far wall max, left internal near wall max and left internal far wall max). These summary variables were then averaged to estimate a single mean-max internal CIMT for each participant visit.
Time Frame: Change from baseline to 36 months
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | 1 Atorvastatin | 2 Placebo
Number analyzed (Participants) | 113 | 108
mm | 0.0090 [0.0052 to 0.0128] | 0.0144 [0.0106 to 0.0182]

6. Secondary Outcome: Change in Mean-Mean Internal CIMT
Description: For the internal carotid arterial segment, mean CIMT values were averaged across angles by side and wall to produce 4 summary variables (right internal near wall mean, right internal far wall mean, left internal near wall mean and left internal far wall mean). These summary variables were then averaged to estimate a single mean-mean internal CIMT for each participant visit.
Time Frame: Change from baseline to 36 months
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | 1 Atorvastatin | 2 Placebo
Number analyzed (Participants) | 113 | 108
mm | 0.0067 [0.0041 to 0.0093] | 0.0082 [0.0056 to 0.0109]

7. Secondary Outcome: Change in Mean-Max Bifurcation CIMT
Description: For each side and wall of the bifurcation arterial segment, the maximum CIMT over the 4 angles of interrogation was selected to produce 4 summary variables (right bifurcation near wall max, right bifurcation far wall max, left bifurcation near wall max and left bifurcation far wall max). These summary variables were then averaged to estimate a single mean-max bifurcation CIMT for each participant visit.
Time Frame: Change from baseline to 36 months
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | 1 Atorvastatin | 2 Placebo
Number analyzed (Participants) | 113 | 108
mm | 0.0033 [0.0001 to 0.0064] | 0.0072 [0.0040 to 0.0104]

8. Secondary Outcome: Change in Mean-Mean Bifurcation CIMT
Description: For the bifurcation arterial segment, mean CIMT values were averaged across angles by side and wall to produce 4 summary variables (right bifurcation near wall mean, right bifurcation far wall mean, left bifurcation near wall mean and left bifurcation far wall mean). These summary variables were then averaged to estimate a single mean-mean bifurcation CIMT for each participant visit.
Time Frame: Change from baseline to 36 months
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | 1 Atorvastatin | 2 Placebo
Number analyzed (Participants) | 113 | 108
mm | 0.0030 [0.0009 to 0.0050] | 0.0055 [0.0035 to 0.0076]

9. Secondary Outcome: Change in Mean-Max Far Wall CIMT
Description: For the far wall measurements for each side and segment, the maximum CIMT over the 4 angles of interrogation was selected to produce 6 summary variables (right common far wall max, right bifurcation far wall max, right internal far wall max, left common far wall max, left bifurcation far wall max, and left internal far wall max). These 6 summary variables were then averaged to estimate a single mean-max far wall CIMT for each participant visit.
Time Frame: Change from baseline to 36 months
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | 1 Atorvastatin | 2 Placebo
Number analyzed (Participants) | 113 | 108
mm | 0.0045 [0.0019 to 0.0072] | 0.0082 [0.0055 to 0.0110]

10. Secondary Outcome: Change in Mean-Mean Far Wall CIMT
Description: For the far wall measurements for each side and segment, mean CIMT values were averaged over the 4 angles of interrogation to produce 6 summary variables (right common far wall mean, right bifurcation far wall mean, right internal far wall mean, left common far wall mean, left bifurcation far wall mean and left internal far wall mean). These 6 summary variables were then averaged to estimate a single mean-mean far wall CIMT for each participant visit.
Time Frame: Change from baseline to 36 months
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | 1 Atorvastatin | 2 Placebo
Number analyzed (Participants) | 113 | 108
mm | 0.0042 [0.0025 to 0.0059] | 0.0064 [0.0047 to 0.0081]

11. Secondary Outcome: Change in Mean-Max Near Wall CIMT
Description: For the near wall measurements for each side and segment, the maximum CIMT over the 4 angles of interrogation was selected to produce 6 summary variables (right common near wall max, right bifurcation near wall max, right internal near wall max, left common near wall max, left bifurcation near wall max, and left internal near wall max). These 6 summary variables were then averaged to estimate a single mean-max near wall CIMT for each participant visit.
Time Frame: Change from baseline to 36 months
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | 1 Atorvastatin | 2 Placebo
Number analyzed (Participants) | 113 | 108
mm | 0.0024 [-0.0003 to 0.005] | 0.0038 [0.0011 to 0.0066]

12. Secondary Outcome: Change in Mean-Mean Near Wall CIMT
Description: For the near wall measurements for each side and segment, mean CIMT values were averaged over the 4 angles of interrogation to produce 6 summary variables (right common near wall mean, right bifurcation near wall mean, right internal near wall mean, left common near wall mean, left bifurcation wall mean and left internal far wall mean). These 6 summary variables were then averaged to estimate a single mean-mean far wall CIMT for each participant visit.
Time Frame: Change from baseline to 36 months
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | 1 Atorvastatin | 2 Placebo
Number analyzed (Participants) | 113 | 108
mm | 0.0022 [0.0002 to 0.0041] | 0.0028 [0.0008 to 0.0047]

13. Secondary Outcome: Change in Natural Log of mg/L for hsCRP
Time Frame: Change from baseline to 36 months
Measure: Mean (95% Confidence Interval); unit: natural log of mg/L
Arm/Group | 1 Atorvastatin | 2 Placebo
Number analyzed (Participants) | 113 | 108
natural log of mg/L | -0.13 [-0.48 to 0.22] | 0.27 [-0.08 to 0.63]

14. Secondary Outcome: Change in Total Cholesterol
Time Frame: Change from baseline to 36 months
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | 1 Atorvastatin | 2 Placebo
Number analyzed (Participants) | 113 | 108
mg/dl | -30.30 [-37.06 to -23.53] | -0.72 [-7.57 to 6.12]

15. Secondary Outcome: Change in HDL Cholesterol
Time Frame: Change from baseline to 36 months
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | 1 Atorvastatin | 2 Placebo
Number analyzed (Participants) | 113 | 108
mg/dl | -0.43 [-2.23 to 1.37] | 0.89 [-0.93 to 2.71]

16. Secondary Outcome: Change in LDL Cholesterol
Time Frame: Change from baseline to 36 months
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | 1 Atorvastatin | 2 Placebo
Number analyzed (Participants) | 113 | 108
mg/dl | -27.63 [-32.79 to -22.47] | -1.48 [-6.72 to 3.76]

17. Secondary Outcome: Change in Triglycerides
Time Frame: Change from baseline to 36 months
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | 1 Atorvastatin | 2 Placebo
Number analyzed (Participants) | 113 | 108
mg/dl | -11.04 [-23.24 to 1.17] | -5.62 [-17.99 to 6.75]

18. Secondary Outcome: Change in Lipoprotein A
Time Frame: Change from baseline to 36 months
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | 1 Atorvastatin | 2 Placebo
Number analyzed (Participants) | 113 | 108
mg/dl | 2.00 [-2.17 to 6.17] | 6.34 [2.09 to 10.59]

19. Secondary Outcome: Change in Homocysteine
Time Frame: Change from baseline to 36 months
Measure: Mean (95% Confidence Interval); unit: μmoles/liter
Arm/Group | 1 Atorvastatin | 2 Placebo
Number analyzed (Participants) | 113 | 108
μmoles/liter | 1.84 [1.08 to 2.60] | 1.76 [0.98 to 2.53]

ADVERSE EVENTS:
Arm/Group | 1 Atorvastatin | 2 Placebo
Serious Adverse Events (participants affected / at risk) | 34/113 | 40/108
Other Adverse Events (participants affected / at risk) | 94/113 | 95/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Atorvastatin (N=113) | 2 Placebo (N=108)
Herpes Zoster (Infections and infestations) | 1 (1) | 5 (5)
Pneumonia (Infections and infestations) | 4 (5) | 1 (5)
Appendicitis (Infections and infestations) | 1 (1) | 1 (2)
Gastroeneritis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Viral Infection (Infections and infestations) | 2 (2) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Cervicitis Trichomonal (Infections and infestations) | 1 (1) | 0 (0)
Clostridial Infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Meningitis Aseptic (Infections and infestations) | 0 (0) | 1 (1)
Meningitis Viral (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis Streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis Acute (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 10 (13) | 8 (10)
Arthraligia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Pscyhotic Disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Drug Dependence (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination, Visual (Psychiatric disorders) | 0 (0) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Lupus Encephalitis (Psychiatric disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Myelitis Transverse (Nervous system disorders) | 0 (0) | 1 (1)
Lupus Nephritis (Renal and urinary disorders) | 1 (1) | 3 (3)
Glomerulonephritis Acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Uticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Panniculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) | 1 (5)
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Adverse Drug Reaction (General disorders) | 1 (1) | 1 (1)
Infusion Related Reaction (General disorders) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Gestational Diabetes (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Abortion, Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Foetal Cardiac Disorder (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 1 (1)
Sickle Cell Anaemia with Crisis (Congenital, familial and genetic disorders) | 1 (5) | 1 (4)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Serum Sickness (Immune system disorders) | 0 (0) | 2 (2)
Histiocytosis haematophagic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Muscle Enzyme Increased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Atorvastatin (N=113) | 2 Placebo (N=108)
Upper Respiratory Tract Infection (Infections and infestations) | 15 (17) | 18 (24)
Sinusitis (Infections and infestations) | 11 (15) | 7 (11)
Urinary Tract Infection (Infections and infestations) | 8 (11) | 10 (16)
Herpes Zoster (Infections and infestations) | 4 (5) | 12 (12)
Bronchitis (Infections and infestations) | 6 (7) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (12) | 10 (15)
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 10 (14) | 8 (11)
Back Pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 5 (5)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 5 (9) | 6 (11)
Myositis (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)
Neurotoxicity (Nervous system disorders) | 27 (62) | 25 (51)
Headache (Nervous system disorders) | 7 (9) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 19 (28) | 28 (47)
Gastrointestinal Disorder (Gastrointestinal disorders) | 10 (14) | 8 (8)
Alanine Aminotransferase Increased (Investigations) | 8 (10) | 9 (11)
Blood Creatine Phosphokinase Increased (Investigations) | 8 (14) | 7 (11)
Aspartate Aminotransferase Increased (Investigations) | 6 (8) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 8 (8)
Non-Cardiac Chest Pain (General disorders) | 6 (7) | 4 (4)
Fatigue (General disorders) | 2 (2) | 6 (6)
Leukopenia (Blood and lymphatic system disorders) | 8 (13) | 6 (9)
Proteinuria (Renal and urinary disorders) | 12 (19) | 8 (11)
Hypertension (Vascular disorders) | 13 (30) | 12 (25)
Conjunctivitis (Eye disorders) | 2 (2) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs agree to follow the CARRA Publication Guidelines. https://www.carragroup.org/about-carra/carra-policies/carra-endorsed-studies-policies